CLINICAL TRIAL: NCT03877159
Title: Analysis of the Variation in Caspase-8 Availability and Cleavage in Oral Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 232080
Record Dates: First submitted 2019-03-11; First posted 2019-03-15 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Other: There is no intervention. — There is no intervention. This is a retrospective study analysing archived tumour samples.

SUMMARY:
Control of cell death is frequently disrupted in cancer resulting in overgrowth of tumour cells. Caspase-8 is a key enzyme involved in controlling cell death. This study examines the importance of caspase-8 in oral cancer.

DETAILED DESCRIPTION:
Control of cell death is frequently disrupted in cancer resulting in overgrowth of tumour cells. The caspase family of enzymes are the key performers of controlled cell death and caspase-8 is frequently mutated in oral cancer. This study will perform DNA sequencing to determine if the gene is wild-type (not mutated). The abundance of inactive (uncleaved) and active (cleaved) caspase-8 will be determined. The levels of the proteins that caspase-8 interacts with (including caspase-3) will be determined. Results will be correlated with tumour stage, patient outcome and the presence of immune cells and other microscopic features. This will improve the understanding of the importance of caspase-8 in oral cancer.

ELIGIBILITY:
Inclusion Criteria:

* Oral cancer
* Sufficient follow up data

Exclusion Criteria:

* Patient has indicated that they do not wish their tissue to be used for research.
* . The quantity or quality of tissue is too little or poor to provide adequate material without significant reserve.
* The material contains bone.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Archived oral cancer tissue specimens within this single institute.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-11-11 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Caspase-8 activity in oral cancer and its impact on disease progression | Up to 3 years
  Molecular analysis of caspase-8 activity will be undertaken and correlated with tumour features and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kennedy, BSc PhD BDS, Principal Investigator — KCL
Locations (1):
- Robert Kennedy, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No patient identifiable data is stored